CLINICAL TRIAL: NCT01729793
Title: A Randomized, Double-Blind, Placebo Controlled, Cross-Over Study to Investigate the Efficacy of Digestive Enzymes on Inflammation After a Meal
Brief Title: Study to Investigate the Efficacy of Digestive Enzymes on Inflammation After a Meal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Enzyme Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NEC-001
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Post Prandial Inflammation Markers
Keywords: TNFalpha; IL6; postprandial; digestive; inflammation; IL1beta; CRP; CBC; ESR
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Digestive Enzyme #2 (Active Comparator): A proprietary blend of dietary supplement enzymes in a capsule
  Interventions: Dietary Supplement: Digestive Enzyme #2
- Placebo (Placebo Comparator): Capsule identical to active arm containing only microcrystalline cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Digestive Enzyme #2 — Contains dietary supplement proteases, lipases and carbohydrases
  Other Names: NEC formula #C372
  Arms: Digestive Enzyme #2
Other: Placebo — Capsule containing microcrystalline cellulose
  Other Names: NEC formula #C373
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the efficacy of Digestive Enzyme Blend #2, a digestive enzyme dietary supplement product, on markers indicative of inflammation after a meal. The markers will be assessed by blood levels tumor necrosis factor alpha (TNF-alpha), interleukin-1 beta (IL-1beta), interleukin-6 (IL-6), and high sensitivity C-reactive protein (hsCRP) at times 0, 45 minutes, 2 hours and 4 hours post-meal. A full complete blood count (CBC)and an erythrocyte sedimentation rate (ESR) blood test will also be conducted at times 0 and 4 hours post-meal. In addition, a questionaire on Gastrointestinal symptoms will be administered 4 hours post-meal. The study hypothesis is that some or all of these potential markers of inflammation will increase following the meal, and the amount of increase in inflammation will be attenuated when a digestive enzyme is consumed with the meal compared to the placebo. In addition, it is hypothesized that levels of gastric discomfort as assessed by the questionaire will be reduced with the digestive enzyme compared to the placebo.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the efficacy of Digestive Enzyme Blend #2, a digestive enzyme dietary supplement product, on markers indicative of inflammation after a meal. The study design is a randomized, double-blind, placebo-controlled, cross-over type study. The markers will be assessed by blood levels TNF-alpha, IL-1beta, IL-6, and hsCRP at times 0, 45 minutes, 2 hours and 4 hours post-meal. A full blood CBC panel and an ESR blood test will also be conducted at times 0 and 4 hours post-meal. In addition, a questionaire on Gastrointestinal symptoms will be administered 4 hours post-meal. The study hypothesis is that some or all of these potential markers of inflammation will increase following the meal, and the amount of increase in inflammation will be attenuated when a digestive enzyme is consumed with the meal compared to the placebo. In addition, it is hypothesized that levels of gastric discomfort as assessed by the questionaire will be reduced with the digestive enzyme compared to the placebo.

ELIGIBILITY:
Inclusion Criteria:

1. If female, not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgical with >1 year since last menstruation). OR Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result.
2. Healthy as determined by laboratory results, medical history and physical exam
3. Agrees to comply with study protocols
4. Has given voluntary, written, informed consent to participate in the study -

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial.
2. Gastrointestinal lesions/ulcer, diabetes, or any condition requiring the use of prescribed medications for treatment
3. Immunocompromised individuals such as subjects that have undergone organ transplantation or subjects diagnosed with human immunodeficiency virus (HIV)
4. History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years after diagnosis are acceptable.
5. History of bleeding disorders, or significant blood loss in the past 3 months
6. Use of blood thinning medications.
7. Use of anti-inflammatory medications, including over-the-counter pain relievers within the past 14 days.
8. Use of prescription medication (other than birth control), vitamins, minerals or other natural health products within the past 3 days. .
9. Alcohol use >2 standard alcoholic drinks per day and/or alcohol or drug abuse within the past year
10. Allergy or sensitivity to study supplement ingredients, study meal ingredients or allergy or sensitivity to yeasts or molds/fungi.
11. Participation in a clinical research trial within 30 days prior to randomization
12. Individuals who are cognitively impaired and/or who are unable to give informed consent
13. Use of fish oil supplements within 10 days of randomization and during the trial
14. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

    -

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
TNF-alpha blood level change from time 0 | 0, 45 minutes, 2 hours and 4 hours
  Aliquots will be taken at time 0 (pre-meal), and the remainder post-meal
IL-1beta blood level change from time 0 | 0, 45 minutes, 2 hours and 4 hours
  Aliquots will be taken at time 0 (pre-meal) and the remainder post-meal.
IL-6 Blood Level change from time 0 | 0, 45 minutes, 2 hours, 4 hours
  Aliquots will be taken at time 0 (pre-meal), and the remainder post-meal
hsCRP Blood Level change from time 0 | 0, 45 minutes, 2 hours, 4 hours
  Aliquots will be taken at time 0 (pre-meal), and the remainder post-meal
CBC Panel change from time 0 | 0, 4 hours
  Aliquots will be taken at time 0 (pre-meal), and the remainder post-meal
ESR blood test change from time 0 | 0, 4 hours
  Aliquots will be taken at time 0 (pre-meal), and the remainder post-meal

SECONDARY OUTCOMES:
Questionaire: Gastrointestinal Symptoms | 4 hours
  The questionaire to assess gastrointestinal symptoms associated with gastrointestinal disturbances will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Study Director — KGK Synergize
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada